CLINICAL TRIAL: NCT03737838
Title: Propagation ANalysis for Arrhythmogenic Conduction Elimination to Prevent Atrial Flutter and Fibrillation
Brief Title: Propagation ANalysis for Arrhythmogenic Conduction Elimination to Prevent Atrial Flutter and Fibrillation (PANACEA-AF)
Acronym: PANACEA-AF
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB17-1769
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Paroxysmal; Atrial; Fibrillation; Ventricular; Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Atrial fibrillation ablation — High density mapping of left atrium using Rhythmia mapping system to identify gaps in conduction and wavefront discontinuities (deceleration zones)

SUMMARY:
The purpose of this study is to perform ultra-high density mapping of the left atrium (a chamber of the heart) using the the Rhythmia Mapping System and to determine whether additional ablation in areas of wavefront discontinuities identified by the map will reduce the likelihood of both atrial fibrillation and atrial flutter.

DETAILED DESCRIPTION:
Catheter ablation (CA) is a class 1 indication for patients with symptomatic drug-refractory atrial fibrillation (AF). With standard pulmonary vein isolation (PVI), the success rate ranges from 60-80% in patients with paroxysmal AF. Despite PVI, certain patients have recurrent AF and often require a repeat ablation procedure.

There is no standard ablation strategy for patients who undergo repeat ablation for recurrent AF. The largest randomized trial to date comparing ablation strategies found that the addition of LA roof and mitral isthmus ablation lines or ablation of LA ganglia was no better than standard PVI. Moreover, the addition of ablation lines in the LA, if not complete, may be pro-arrhythmic and lead to the development of LA AFL, which is often more symptomatic that AF itself.

Ultra-high density mapping during sinus rhythm allows for rapid creation of isochronal late activation maps (ILAM) in patients with ventricular tachycardia. To date, creating ILAM of the LA has not been reported and it is not known whether additional ablation in these areas improves freedom from all atrial tachyarrhythmias at 1 year follow-up. Moreover, ablation at the deceleration zones and/or gaps identified using ultra-high density mapping is a promising strategy to improve ablation success and decrease the potential for recurrent AF.

The rationale of the study is two-fold.

1. This study would be the first to report ILAM in the LA and confirm that the diseased LA may behave similarly to the diseased left or right ventricle.
2. Ablation of gaps and/or deceleration zones in the LA would be a novel approach to treat patients with recurrent AF after initial PVI, and if successful, provide another strategy to treat these refractory problems.

Co-PIs:

Hemal Nayak, MD Guarav Upadhyay, MD Andrew Beaser, MD Zaid Aziz, MD

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Re-do AF ablation with history of PVI
* Undergone at least 1 prior ablation

Exclusion Criteria:

* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Recent stroke within 6 months of planned procedure
* Inability to take oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of patients with AF refractory to prior ablation
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Freedom from recurrent atrial fibrillation and atrial flutter | Baseline to 1 year
  Freedom from atrial arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Tung, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anter E, Tschabrunn CM, Buxton AE, Josephson ME. High-Resolution Mapping of Postinfarction Reentrant Ventricular Tachycardia: Electrophysiological Characterization of the Circuit. Circulation. 2016 Jul 26;134(4):314-27. doi: 10.1161/CIRCULATIONAHA.116.021955. PMID 27440005
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Irie T, Yu R, Bradfield JS, Vaseghi M, Buch EF, Ajijola O, Macias C, Fujimura O, Mandapati R, Boyle NG, Shivkumar K, Tung R. Relationship between sinus rhythm late activation zones and critical sites for scar-related ventricular tachycardia: systematic analysis of isochronal late activation mapping. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):390-9. doi: 10.1161/CIRCEP.114.002637. Epub 2015 Mar 4. PMID 25740836
- [Background] Anter E, McElderry TH, Contreras-Valdes FM, Li J, Tung P, Leshem E, Haffajee CI, Nakagawa H, Josephson ME. Evaluation of a novel high-resolution mapping technology for ablation of recurrent scar-related atrial tachycardias. Heart Rhythm. 2016 Oct;13(10):2048-55. doi: 10.1016/j.hrthm.2016.05.029. Epub 2016 Jun 1. PMID 27262767
- [Background] Viswanathan K, Mantziari L, Butcher C, Hodkinson E, Lim E, Khan H, Panikker S, Haldar S, Jarman JW, Jones DG, Hussain W, Foran JP, Markides V, Wong T. Evaluation of a novel high-resolution mapping system for catheter ablation of ventricular arrhythmias. Heart Rhythm. 2017 Feb;14(2):176-183. doi: 10.1016/j.hrthm.2016.11.018. Epub 2016 Nov 17. PMID 27867071
- [Background] Luther V, Sikkel M, Bennett N, Guerrero F, Leong K, Qureshi N, Ng FS, Hayat SA, Sohaib SM, Malcolme-Lawes L, Lim E, Wright I, Koa-Wing M, Lefroy DC, Linton NW, Whinnett Z, Kanagaratnam P, Davies DW, Peters NS, Lim PB. Visualizing Localized Reentry With Ultra-High Density Mapping in Iatrogenic Atrial Tachycardia: Beware Pseudo-Reentry. Circ Arrhythm Electrophysiol. 2017 Apr;10(4):e004724. doi: 10.1161/CIRCEP.116.004724. PMID 28356307
- [Background] Ciaccio EJ, Chow AW, Davies DW, Wit AL, Peters NS. Localization of the isthmus in reentrant circuits by analysis of electrograms derived from clinical noncontact mapping during sinus rhythm and ventricular tachycardia. J Cardiovasc Electrophysiol. 2004 Jan;15(1):27-36. doi: 10.1046/j.1540-8167.2004.03134.x. PMID 15028069
- [Background] Anter E, Tschabrunn CM, Contreras-Valdes FM, Li J, Josephson ME. Pulmonary vein isolation using the Rhythmia mapping system: Verification of intracardiac signals using the Orion mini-basket catheter. Heart Rhythm. 2015 Sep;12(9):1927-34. doi: 10.1016/j.hrthm.2015.05.019. Epub 2015 May 19. PMID 26001505
- [Background] Wann LS, Curtis AB, January CT, Ellenbogen KA, Lowe JE, Estes NA 3rd, Page RL, Ezekowitz MD, Slotwiner DJ, Jackman WM, Stevenson WG, Tracy CM; 2011 Writing Group Members; Fuster V, Ryden LE, Cannom DS, Le Heuzey JY, Crijns HJ, Lowe JE, Curtis AB, Olsson S, Ellenbogen KA, Prystowsky EN, Halperin JL, Tamargo JL, Kay GN, Wann L; 2006 Writing Committee Members; Jacobs AK, Anderson JL, Albert N, Hochman JS, Buller CE, Kushner FG, Creager MA, Ohman EM, Ettinger SM, Stevenson WG, Guyton RA, Tarkington LG, Halperin JL, Yancy CW; ACCF/AHA Task Force Members. 2011 ACCF/AHA/HRS focused update on the management of patients with atrial fibrillation (updating the 2006 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Jan 4;123(1):104-23. doi: 10.1161/CIR.0b013e3181fa3cf4. Epub 2010 Dec 20. No abstract available. PMID 21173346